CLINICAL TRIAL: NCT03485963
Title: A Phase I Study to Evaluate the Safety, Immunologic, and Virologic RESponses of HIV-Specific T-cells With Non-escaped Epitope Targeting (HST-NEETs) as a Therapeutic Strategy in HIV-Infected Individuals on Antiretroviral Therapy During Acute And Chronic Infection
Brief Title: HIV-1 Specific T -Cells (HST-NEETs) for HIV-Infected Individuals
Acronym: RESIST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director, center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009968
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fixed dose HIV-1 specific T-cells (HST-NEETs) (Experimental): Patients will be screened for eligibility in Step 1 and undergo a blood draw of 100-120mL to allow production of autologous HST-NEETS. patients will receive a fixed dose of 2x10e7/m2. For the first 3 recipients, the infusions will occur 4 weeks apart. If no adverse reactions occur that are attributable to the HST-NEETs, the recipients thereafter will receive the two infusions separated by 2 weeks.
  Interventions: Biological: HST-NEETs

INTERVENTIONS:
Biological: HST-NEETs — The primary objective of this study is to evaluate the safety and tolerability of expanded HIV-specific T cell therapy (HST-NEETs) in HIV-infected individuals suppressed on cART. Patients with a partial response or stable disease 8 weeks after T-cell infusion were eligible to receive additional T-cells, consisting of the same number of cells as their second injection.

SUMMARY:
This is a phase I, multi-site, study of the safety, immunologic and virologic responses of ex vivo expanded HIV-1 multi-antigen specific T-cell therapy (HST-NEET) as a therapeutic strategy in HIV-infected individuals suppressed on antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Treatment Description: This is a phase I, multi-site, study of the safety, immunologic and virologic responses of ex vivo expanded HIV-1 multi-antigen specific T-cell therapy (HST-NEET) as a therapeutic strategy in HIV-infected individuals suppressed on ART. Patients will be screened for eligibility in Step 1 and undergo a blood draw of 100-120mL to allow production of autologous HST-NEETS. Those meeting study eligibility and with successful production of HST-NEETs will then enter Step 2 where patients have the OPTION of being enrolled on a separate GWU Protocol 04216 to obtain a pre- and post- HST-NEET treatment leukapheresis procedure to measure the frequency of HIV-1 infection of resting CD4+ T cells using the viral outgrowth assay. All participants will then receive (within 30 days of the leukapheresis procedure if applicable) the same treatment and dose (2x107/m2) of HST-NEETs in Step 2. For the first 3 recipients, the infusions will occur 4 weeks apart. If no adverse reactions occur that are attributable to the HST-NEETs, the recipients thereafter will receive the two infusions separated by 2 weeks.

Sample Size and Study Duration: Up to 12 HIV-infected individuals followed for 48 weeks.

Accrual Objective: The total sample size is 12 participants. Participants will be followed for 48 weeks. Because the focus of the study is on safety and potential adverse events are most likely to occur within 28 days of administration, accrual will be staggered such that enrollment and treatment administration will include a maximum of 1 participant per week. Participants who do not receive study treatment will be replaced. In addition, any participant who is not administered the full study treatment infusion, or discontinues the study prior to day 28 without having met the primary safety endpoint will be replaced until the target enrollment of participants is met.

ELIGIBILITY:
Inclusion Criteria:

Recipient Inclusion Criteria for cell procurement and cell infusion:

* ≥ 18 years and < 65 years of age
* Confirmation of HIV-1 infection

  - any licensed ELISA test kit which is confirmed by Western blot or Multispot HIV-1/HIV-2 assay prior to screening. HIV culture, HIV antigen, plasma HIV RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* On potent antiretroviral therapy, defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor without interruption (Interruption is defined as missing doses by self report for no more than two (2) consecutive days or more than four (4) cumulative days) in the 12 weeks prior to cell procurement for HST NEETs manufacturing. Other potent fully suppressive antiretroviral combinations will be considered on a case- by-case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, toxicity, or other reasons are permitted if an alternative suppressive regimen was maintained under the compliance criteria above.
* Stable ART regimen for minimum of 12 weeks with no detectable HIV RNA concentrations as defined above. Participants may have had one or more changes in their ART regimen during the 12 week for tolerance, or dosing simplification.
* Ability and willingness of participant to continue and be compliant with cART throughout the study.
* Plasma HIV-1 RNA below detectable limit by conventional CLIA approved assays (<50 copies/mL) for ≥ 1 year. A single unconfirmed plasma HIV RNA > limit of detection but < 1000 c/mL is allowed within the 12 months prior to screening/cell donation but none in the preceding 6 months, is permitted provided that a repeat RNA was < 20.
* Plasma HIV-1 RNA < 50 copies/mL at screening.
* CD4+ cell count > 350 cells/mm3 at screening.
* Karnofsky score of ≥ 50%
* No active HCV infection (measureable HCV RNA) within 90 days of cell procurement.
* No active HBV infection (measureable HBV DNA or HBVsAg+) within 90 days of cell procurement.
* All female participants participating in sexual activity that could lead to pregnancy must agree to use at least two of the following reliable methods of birth control (at least one of which is a barrier method) for at least 21 days prior to study entry, continuing and until 12 weeks after the last dose of the study product: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, Intrauterine Device, hormone-based contraceptive, tubal ligation, NuvaRing.
* All male participants participating in sexual activity that could lead to pregnancy must agree to use condoms for at least 21 days prior to study entry, continuing and until 12 weeks after the last dose of the study product.
* Ability and willingness of subject to give written informed consent.
* Ability and willingness to provide adequate locator information and contact information for at least 2 adults who can reach the participant within 24 hours
* Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
* Adequate vascular access (peripheral and central) for HST-NEET infusion.

Exclusion Criteria:

* Prior use of any HIV immunotherapy or vaccine within 12 months prior to Screening.
* Use of any of the following within 90 days prior to entry: immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, IFN, interleukin-2 (IL-2), Coumadin, warfarin, or other Coumadin derivative anticoagulants.
* Patients on a CCR5 inhibitor or an entry inhibitor are not eligible for participation in the study
* Received any infusion blood product, immune globulin, or hematopoietic growth factors within 90 days prior to study entry.
* History of malignancy, immunodeficiency other than HIV, or any other condition that would make the subject unsuitable for the study in the opinion of the performance site PIs.
* Any active malignancy that may require chemotherapy or radiation therapy.
* Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) within 4 weeks prior to study entry.
* Inability to comply with study requirements, which could impact study integrity and/or safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Product-Emergent Adverse Events | from the first day of study treatment until 28 days after the last infusion.
  Occurrence of any ≥ Grade 3 AE including signs/symptoms, lab toxicities, and/or clinical events, that is possibly, probably or definitely related to study treatment any time from the first day of study treatment until 28 days after the last infusion. Safety data will include local and systemic signs and symptoms, laboratory measures of safety/toxicity, and all adverse and serious adverse events. Safety data will be routinely collected throughout the duration of the study. Relationship to study treatment will be judged by the protocol team. If any Grade 4 or 5 Serious Adverse Events occur, this will trigger an immediate pause in the protocol while the relationship to the T cell therapeutic is evaluated. If the attribution is deemed probably or definitely related to the study agent, the protocol will stop.

SECONDARY OUTCOMES:
HST-NEETS responses | 12 months
  Determine the number of patients who respond to HST_NEETS

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keller, MD, Principal Investigator — CNMC
Locations (3):
- United States (3):
  - Whitman Walker Health Research Department (Wwh), Washington D.C., District of Columbia
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center and WHITMAN WALKER HEALTH RESEARCH DEPARTMENT (WWH), Washington D.C., District of Columbia